CLINICAL TRIAL: NCT06149741
Title: Defunctioning Left-sided Colostomy in Low Anterior Resection for Rectal Cancer
Acronym: STOMALEFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Collaborators: Sunderby Hospital (Other); Östersund Hospital (Unknown); Sundsvall Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UmU-STOMALEFT
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Left-sided loop colostomy (Experimental): Left-sided loop colostomy matured in left iliac fossa after complete splenic flexure mobilisation, mesorectal excision and anastomosis
  Interventions: Procedure: Defunctioning left-sided loop colostomy

INTERVENTIONS:
Procedure: Defunctioning left-sided loop colostomy — Descending or left transverse double-barrelled loop colostomy in left iliac fossa after complete splenic flexure mobilisation, mesorectal excision, and anastomosis.

SUMMARY:
This is prospective, multi centre study evaluating a novel type of defunctioning loop stoma after low anterior resection for rectal cancer. Patients will be operated with a complete splenic flexure mobilisation and total mesorectal excision. An anastomosis will be fashioned at the pelvic floor. This will leave a redundant colon which will be brought up and matured in the left iliac fossa. Patient bowel function and quality of life will be monitored at baseline and at one year postoperatively, when the stoma will typically have been reversed. Dehydration and kidney injury are expected to become infrequent in comparison with the main alternative loop ileostomy. About 20 patients will be included in this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Capacity for informed consent
* Planned defunctioning stoma
* Planned mesorectal excision with anastomosis for rectal cancer

Exclusion Criteria:

* Manifest atherosclerotic disease (peripheral vascular disease, previous myocardial infarction, angina, etc)
* Previous oncological colonic resection
* Defunctioning stoma in situ
* Intraoperative event leading to bowel resection and subsequent inability to bring out left-sided colostomy without tension on the anastomosis
* Intraoperative circumstances as judged by the operating surgeon leading to unacceptable risks due to loop colostomy placement (abdominal wall size, short mesentery, other preconditions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Low anterior resection syndrome (LARS) | 1 year
  Rate of major LARS (score 31-42) as measured by the LARS questionnaire, which assesses bowel dysfunction.

SECONDARY OUTCOMES:
Bowel ischaemia | 30 days
  Rate of ischaemia/necrosis of the colonic limb due to marginal artery compromise.

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå University Hospital, Umeå, Sweden